CLINICAL TRIAL: NCT03311893
Title: the Rate of Awareness and Acceptability of Natural Orifice Surgeon in Middle Eastern Society is Similar to Other Studies
Brief Title: Determine the Point of View of Society Society to Natural Orifice Surgeon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ersin Gündoğan, operator doctor, Inonu University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016/199
Record Dates: First submitted 2017-09-13; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2016-10

CONDITIONS: Health, Subjective
MeSH Terms: interventions — Natural Orifice Endoscopic Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health personnel (Active Comparator): natural orifice surgery evaluation of the awareness of the use of transvaginal, transoral and trananal approach in surgical excision and the difference between the health staff and population
  Interventions: Procedure: natural orifice surgery
- population (Placebo Comparator): natural orifice surgery evaluation of the awareness of the use of transvaginal, transoral and trananal approach in surgical excision and the difference between the health staff and population
  Interventions: Procedure: natural orifice surgery

INTERVENTIONS:
Procedure: natural orifice surgery — evaluation of the awareness of the use of transvaginal, transoral and transcranial approach in surgical excision and the difference between the health staff and the pathology

SUMMARY:
200 participants' perception and acceptability of natural hole surgeon

DETAILED DESCRIPTION:
100 participants health personnel 100 participants population two group's perception and acceptability of natural orifice surgeon

ELIGIBILITY:
Inclusion Criteria:

* all female (health personnel and population)

Exclusion Criteria:

* none

Ages: 17 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
natural orifice surgery | 12 months
  a survey study that measures the awareness of natural orifice surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ersin Gündoğan, MD, Principal Investigator — Inonu Unıversity- general surgery

IPD SHARING:
Plan to Share IPD: Undecided